CLINICAL TRIAL: NCT06246760
Title: Prestación de Servicios científicos, evaluación y Control Del Rendimiento
Brief Title: Differences in Ventilatory Function, Body Composition, and Cardiorrespiratory Fitness According to Training Status
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, ANA BELEN PEINADO LOZANO, Principal Investigator, Universidad Politecnica de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PSC191100471
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Body Composition; Cardiovascular Health; Ventilatory Physiology
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Incremental exercise test (Experimental): Maximal incremental exercise test on a treadmill or a cycle ergometer until volitional exhaustion
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Incremental exercise test until volitional exhaustion

SUMMARY:
The goal of this cross-over study is to evaluate the physiological response to exercise and body composition according to training status in participants with a wide spectrum of fitness states. The main questions it aims to answer are:

* Which are the physiological differences across participants with different training status?
* Which are the body composition differences across participants with different training status?

DETAILED DESCRIPTION:
To satisfy the objective of the project, participants will perform an incremental test until volitional exhaustion. During this test, respiratory gases will be measured via a gas analyser as well as the cardiac response via an electrocardiogram. The same participants will have their body composition measured by dual X-ray densitometry (DXA).

ELIGIBILITY:
Inclusion Criteria:

* Be in enough physical fitness to perform the incremental test to volitional exhaustion.

Exclusion Criteria:

* Present any health condition preventing to perform the incremental exercise test until volitional exhaustion.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1272 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Training status | breath-by-breath during the whole test
  Oxygen uptake at ventilatory threshold 1, ventilatory threshold 2 and maximal oxygen uptake
Body composition | one determination before the test
  Fat mass (kg), fat free mass (kg), fat mass percentage, fat-free mass (FFM) percentage, weight (kg), and height (m). These variables are assesed by dual-energy X-ray absorptiometry (DXA).
Bone mineral density | one determination before the test
  Total, lumbar spine and femoral neck bone mineral density (g/cm^2). These variables are assesed by dual-energy X-ray absorptiometry (DXA).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical activity and sport sciences, Madrid, Comunity of Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
In accordance with the law 15/1999 on the protection of personal data, the personal data required are those necessary for scientific purposes, for possible studies that may be carried out. In none of these possible studies will your name appear and your identity will not be revealed to any person except to fulfil the purposes of the study, and in the event of a medical emergency or legal requirement. Any personally identifiable information will be retained and processed under secure conditions for the purpose of determining the results of possible studies. The results of these studies may be communicated to health authorities and the scientific community through conferences and/or publications.

REFERENCES:
- [Derived] Benitez-Munoz JA, Alcocer-Ayuga M, Cupeiro R, Guisado-Cuadrado I, Rojo-Tirado MA, Alfaro-Magallanes VM, Romero-Parra N, Aparecida-Castro E, Ramos-Campo DJ, Armero-Sotillo A, Peinado AB, Benito PJ. Ventilatory Thresholds Differences According to Aerobic Fitness Level in 1450 Males and 241 Females on Cycle-Ergometer: A Cross-Sectional Study. Eur J Sport Sci. 2025 Jul;25(7):e12323. doi: 10.1002/ejsc.12323. PMID 40528561
- [Derived] Benitez-Munoz JA, Benito PJ, Guisado-Cuadrado I, Cupeiro R, Peinado AB. Differences in the ventilatory thresholds in treadmill according to training status in 971 males and 301 females: a cross-sectional study. Eur J Appl Physiol. 2025 Feb;125(2):499-510. doi: 10.1007/s00421-024-05622-z. Epub 2024 Sep 24. PMID 39316126